CLINICAL TRIAL: NCT02682953
Title: Hyperbaric Oxygen Therapy for Hematopoietic Progenitor Cell Collection in Poor Mobilizers
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: subject recruitment not feasible due to standard care changes
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: Healogics (Unknown)
Responsible Party: Principal Investigator, Stephen Thom, Professor, University of Maryland, Baltimore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HP-00064099
Record Dates: First submitted 2016-02-09; First posted 2016-02-17 (Estimated); Last update posted 2019-12-11 (Actual); Status verified 2019-12

CONDITIONS: Bone Marrow Transplantation; Hematopoietic Stem Cells; Multiple Myeloma; Lymphoma
MeSH Terms: conditions — Multiple Myeloma; Lymphoma | interventions — Filgrastim; plerixafor; Hyperbaric Oxygenation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Hyperbaric oxygen therapy (Experimental): Exposure to oxygen at 2.4 atmospheres absolute for 90 minutes/day for 3 to 5 days
  Interventions: Drug: Neupogen; Procedure: Hyperbaric oxygen therapy; Drug: Plerixafor

INTERVENTIONS:
Drug: Neupogen — Pharmacological agents often used for stem cell mobilization will be utilized in this study.
  Other Names: Plerixafor
Procedure: Hyperbaric oxygen therapy — Exposure to oxygen at 2.4 atmospheres absolute for 90 minutes/day for 3 to 5 days
Drug: Plerixafor — Pharmacological agents often used for stem cell mobilization will be utilized in this study.

SUMMARY:
This is a pilot study to evaluate the efficacy of hyperbaric oxygen therapy (HBO2) for mobilizing hematopoietic progenitor cells from bone marrow to blood. These cells are needed for patients to undergo bone marrow transplantation and some patients fail to respond to current best chemotherapy. HBO2 has been shown to trigger stem cell mobilization in other patient populations and we plan to investigate whether this intervention can act in concert with chemotherapeutic agents to allow poor mobilizer patients to achieve successful bone marrow transplantation. Twenty patients will be identified by participating hematologists who have failed to respond adequately to chemotherapy. When it is deemed appropriate to attempt an additional stem cell mobilization protocol, these patients will be administered chemotherapy as determined by their primary treating hematologist and additionally receive daily HBO2 (2.5 atmospheres absolute [ATA] for 90 minutes) for 3-8 days. At intervals, blood samples will be obtained as is the normal transplantation protocol practice to assess whether adequate stem cells are present in blood for the patient to proceed with transplantation. The project is anticipated to take one year to complete.

DETAILED DESCRIPTION:
Study subjects will be patients who have failed to achieve an adequate mobilization of hematopoietic progenitor cells (so-called stem cells) into their blood stream to safely proceed with hematopoietic stem cell transplantation as a component of treatment for a hematological malignancy. There are several possible chemo-mobilization procedures that a primary clinician may prescribe and when blood cell counts at the end of these procedures document an inadequate number for transplantation, there is no accepted clinical course of action other than to repeat the procedures and sometimes add another drug, such as plerixafor. This investigation is based on a single center abstract presented at a hematological meeting (the 2012 ASCO University Annual Meeting) where 7 of 9 patients previously identified as poor mobilizers achieved sufficient mobilization with addition of hyperbaric oxygen therapy to standard care (1). This project is to recapitulate the study in a somewhat larger patient population (20 subjects).

Once an individual has been identified as a poor mobilizer, meaning they failed with standard therapy to mobilize sufficient stem cells to proceed with bone marrow transplantation, they will be approached by one of the investigators, informed of the study and asked to sign informed consent. After a period of time identified as a 'rest period' (typically 2-4 weeks, exact duration is a decision to be made by the primary clinician overseeing the patient's care) they will begin treatment in another attempt to mobilize an adequate number of hematopoietic progenitor cells (defined as 2 x 10^6 cells/kg body weight). A blood sample will be obtained to determine the baseline number of stem cells (an aspect of normal clinical care) and also an extra 4 ml tube of blood will be obtained for additional studies to be done in the PI's lab (these are added evaluations of hypoxia inducible factors (HIF) within circulating stem cells that may influence function but are not currently recognized as having clinical relevance).

A component of normal care at this point is daily injections with a drug called Neupogen. In order to accommodate the needed time for normal clinical procedures with the anticipated time-course for hyperbaric oxygen therapy-induced stem cell mobilization, the study protocol will begin on Thursday with Neupogen injection plus a 90 minute exposure to hyperbaric oxygen at a pressure of 2.4 atmospheres absolute (the normal protocol followed by the Hyperbaric Oxygen [HBO2] Therapy Service for daily treatments of elective patients). Neupogen plus HBO2 will be repeated again on Friday, and on Saturday and Sunday Neupogen injections again administered.

On Monday Neupogen plus HBO2 will be repeated and on Tuesday morning a blood sample will be obtained. This is for counting stem cells to asses if an adequate number is mobilized (hence an aspect of normal clinical care) and also an extra 4 ml tube of blood will be obtained for the additional studies of HIF in stem cells to be done in the PI's lab. If the cell count exceeds 20/ml blood the subject will undergo apheresis to harvest stem cells on that day. If the cell count is less than 20/ml, the subject will again receive a Neupogen injection and HBO2 and an additional drug that is part of normal care called plerixafor. On Wednesday morning a blood sample will again be obtained to asses if an adequate stem cell number is mobilized (hence an aspect of normal clinical care) and also an extra 4 ml tube of blood will be obtained for additional studies to be done in the PI's lab. If the cell count exceeds 20/ml blood the subject will undergo apheresis to harvest stem cells on that day. If the cell count is still less than 20/ml blood, the subject will again receive a Neupogen injection and HBO2 and an additional dose of plerixafor. It is anticipated that by Thursday morning, when another blood cell count will be done, the study subject will be able to proceed with harvesting their stem cells by the apheresis procedure.

Doses and agents used for chemotherapy will be determined by a patient's primary treating hematologist according to standard treatment guidelines (Neupogen and plerixafor). The experimental intervention will be inclusion of daily HBO2 (2.4 ATA for 90 minutes) administered for 3-5 days. Assessment of blood progenitor cell mobilization will follow standard clinical evaluations and protocols. No additional interventions will be performed. The only addition to standard clinical analysis will be obtaining an extra 4 ml tube of blood at each phlebotomy session for studies to be performed in the PI's lab including analysis of progenitor cell sub-types, content of hypoxia inducible factors and activity of nitric oxide synthase-3 in platelets following published methods (3).

ELIGIBILITY:
Inclusion Criteria:

1. Clinical indication for hematopoietic stem cell transplantation.
2. Those failing to achieve an adequate collection of progenitor cells with standard chemotherapy treatment to safely perform hematopoietic stem cell transplantation.

Exclusion Criteria:

1. Diabetes mellitus
2. Renal or other organ transplantation and on immunosuppressive agents
3. NYHA Class III or IV heart failure
4. Liver cirrhosis
5. HIV infection and/or AIDS
6. Seizure disorder and not taking anti-seizure medications
7. Asthma/bronchospasm not resolvable with inhaled bronchodilators
8. Eustachian tube dysfunction and inability to equalization of pressure across the middle ears
9. Confinement anxiety not controlled with oral benzodiazepine therapy.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-10; Primary Completion 2017-02 (Estimated); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Number of patients who adequately mobilize stem cells to undergo bone marrow transplantation. | 1-2 years
  Among entered patients, the number who adequately mobilization of stem cells to proceed with bone marrow transplantation

CONTACTS AND LOCATIONS:
Locations (1):
- University of Maryland Medical Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Data on stem cell changes with treatment